CLINICAL TRIAL: NCT01394094
Title: Effects of Gum Chewing on Recovery of Bowel Function Following Benign Gynecologic Surgery: a Randomized Controlled Trial
Brief Title: Effects of Gum Chewing on Recovery of Bowel Function Following Benign Gynecologic Surgery
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chiang Mai University (Other)
Responsible Party: Manatsawee Manopunya, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 10OCT010402
Record Dates: First submitted 2011-07-13; First posted 2011-07-14 (Estimated); Last update posted 2011-07-14 (Estimated); Status verified 2011-07

CONDITIONS: Recovery of Bowel Function, Due to Gum Chewing
Keywords: Gum chewing; Bowel function; benign gynecologic surgery
MeSH Terms: interventions — Chewing Gum

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gum Chewing (Experimental): Gum chewing (30 minutes in duration each time, 4 times/days at the usual time of meal, until the first flatus) in addition to conventional postoperative feeding schedule
  Interventions: Behavioral: Gum chewing
- Conventional (No Intervention): Conventional postoperative feeding schedule

INTERVENTIONS:
Behavioral: Gum chewing — Gum chewing(30 minutes in duration each time, 4 times/days at the usual time of meal, until the first flatus) in the addition to conventional postoperative feeding schedule
  Other Names: Sugar free and calcium free gum
  Arms: Gum Chewing

SUMMARY:
Gum chewing can promotes the return bowel function after gynecologic surgery.

DETAILED DESCRIPTION:
Following abdominal surgery for treatment of benign gynecologic surgery, paralytic ileus may be develops. Gum chewing can promotes the return of bowel function through the cephalic-vagal reflex and increased intestinal enzymes secretion. This study will be evaluate effects of adding gum chewing to the conventional postoperative feeding protocol on the return of bowel function, its related complication, and patients's satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing abdominal surgery for benign gynecologic conditions at Maharaj Nakorn Chiang Mai hospital

Exclusion Criteria:

* Perioperative hyperalimentation
* Recent chemotherapy (within 3 weeks before surgery)
* Previous bowel surgery
* Inflammatory bowel disease
* Previous abdominal or pelvic radiation
* Need for immediate postoperative endotracheal intubation
* Need for postoperative admission to intensive care unit
* Undergoing emergency surgery with oral intake of fluid or food with in 4 hours before surgery

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2011-07; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Time to first flatus | Up to 7 days after surgery

SECONDARY OUTCOMES:
Incidence and severity of postoperative nausea, vomiting and abdominal discomfort | Up to 7 days after surgery
Incidence of postoperative complications | Up to 7 days after surgery
Time to first regular diet | Up to 7 days after surgery
Time to first defecation | Up to 7 days after surgery
Hospital stay | Up to 7 days after surgery
Patients's satisfaction | Up to 7 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Manatsawee - Manopunya, MD, Principal Investigator — Chiang Mai University, Thailand
Locations (1):
- Faculty of Medicine, Chiang Mai University, Amphoe Muang, Chiang Mai, Thailand